CLINICAL TRIAL: NCT05162547
Title: Multi-Center Clinical Performance Evaluation of the NeuMoDx™ FluA/FluB/RSV/Severe Acute Respiratory Syndrome-CoV-2 Assay on the NeuMoDx™ Molecular Systems
Brief Title: Clinical Performance Evaluation of the NeuMoDx™ FluA/FluB/RSV/Severe Acute Respiratory Syndrome-CoV-2 Assay
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SMF-21-2526-0-001
Record Dates: First submitted 2021-12-09; First posted 2021-12-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh and frozen leftover specimens from nasopharyngeal (NP) specimens collected from symptomatic individuals in transport medium.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: NeuMoDx™ FluA/FluB/RSV/SARS-CoV-2 Assay — The NeuMoDx™ FluA/FluB/RSV/SARS-CoV-2 Assay (IUO) is a multiplexed, in vitro real-time Polymerase Chain Reaction assay, diagnostic test intended for the simultaneous qualitative detection and differentiation of Influenza A virus (Flu A), Influenza B virus (Flu B), Respiratory Syncytial Virus (RSV) and SARS-CoV-2 RNA

SUMMARY:
To demonstrate the clinical performance of the NeuMoDx™ FluA/FluB/RSV/SARS-CoV-2 Assay on the NeuMoDx Systems by determining clinical sensitivity and specificity of the Assay.

DETAILED DESCRIPTION:
To evaluate the clinical performance of the NeuMoDx™ FluA/FluB/RSV/SARS-CoV-2 Assay on the on the NeuMoDx™ 288 and 96 Molecular Systems, collectively referred to as NeuMoDx Systems. The results of this study will be used to support regulatory registration and product release in the US, Europe and other markets.

ELIGIBILITY:
Inclusion Criteria:

* Fresh specimens shall be collected from all comers across the study duration
* Collected from individuals of any age presenting with influenza-like illness (ILI)
* Nasopharyngeal (NP) swab specimen obtained using a flexible mini-tip flocked swab and collected into 3 mL Copan® Universal Transport Media (UTM) [Cat. No.305c] or Beckton Dickinson (BD™) Universal Viral Transport (UVT) [Cat. No. 220531]
* Minimum volume for residual specimen approximately 2 mL
* Fresh specimens to be tested within 3 days of collection.
* Fresh specimens to be stored under the recommended stability conditions (2-8°C).

Exclusion Criteria:

* Required information unable to be obtained from associated medical chart.
* Specimens not fitting criteria outlined above.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals presenting with influenza-like illness from all age groups
Sampling Method: Probability Sample
Enrollment: 2383 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Positive Percentage Agreement | 6 months
  positive percentage agreement

SECONDARY OUTCOMES:
Negative Percentage Agreement | 6 months
  negative percentage agreement

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — QIAGEN Gaithersburg, Inc
Locations (1):
- QIAGEN Gaithersburg, Inc, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
all samples are residual and anonymized